CLINICAL TRIAL: NCT04427358
Title: RT-PCR SARS-CoV-2 at 1 Month of COVID-19 Infection in the Geriatric Population
Acronym: COVID-19GAOM
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7838
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-06

CONDITIONS: Covid-19
Keywords: RT-PCR SARS-CoV-2; Covid-19; Carriage; Viral shredding; Elderly; Elderly people; Geriatric
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the rate of positive RT-PCR SARS-CoV-2 test at 1 month of COVID infection among elderly people.

It is unclear how long an individual with COVID-19 will remain "sick" and "contagious". It appears that SARS-CoV-2 can be transmitted before symptoms appear and throughout the course of the disease.

They investigators did not find any study on a COVID + geriatric population reassessing carriage at 1 month even though age seems to be a risk factor for prolonged excretion as suggested in the study following study: Xu K, Chen Y, Yuan J, Yi P, Ding C, Wu W, et al. Factors associated with prolonged viral RNA shedding in patients with COVID-19. Clinical Infectious Diseases. 2020 Apr 9; ciaa351

ELIGIBILITY:
Inclusion Criteria:

* Age> 70years
* Patient hospitalized on the geriatric center from March 1, 2020 to August 1, 2020 with a diagnosis of COVID-19 still alive at 1 month.
* Patient having agreed to the re-use of their data for the purposes of this research

Exclusion Criteria:

* Subject who expressed his opposition to participate in the study
* Subject under judicial protection

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Patient over 70 years age having COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
1. Analysis of the rate of RT-PCR SARS-CoV-2 positive at 1 month of COVID infection | at 1 month of COVID infection]
2. Assess quantitative evaluation of a nasopharyngeal swab SARS-CoV-2 RT-PCR test | at 1 month after COVID infection
  The objective of this study is to quantitatively assess viral shedding in COVID-19 infected elderly patients who survived infection in order to provide an overview of the evolution of nasopharyngeal swab SARS-CoV-2 real-time reverse transcriptase-polymerase chain reaction (RT-PCR) test results with the Cycle threshold value of the RT-PCR test.. The investigatrors analyze nasopharyngeal RT-PCR at diagnosis. After one month since the date of onset symptoms they reassessed survival patients with nasopharyngeal RT-PCR and repeat the RT-PCR at least every week until final negative conversion occurs.

SECONDARY OUTCOMES:
Assessment of late stool SARS-CoV-2 RT-PCR, serological status and associated factors with death and RT-PCR results 1 month after the date of first symptom onset | 1 month after the date of first symptom onset
  * Assessment of late stool SARS-CoV-2 RT-PCR results one month after the date of onset symptom(dso) (% of patients with a positive fecal RT-PCR test after 1 month)
  * COVID-19 serological status; associated factors with death and RT-PCR results 1 month after the dso: Age (year), gender, Medical history prior to hospilization : Hypertension, diabetes, coronary artery disease, heart failure, atrial fibrillation, chronic respiratory disease, History of medication: ACEI, ARBs Antiplatetet drug, doses of anticoagulant therapy, antibiotic, corticotherapy, statin, Proton pump inhibitor, T°C>37.8 7 days after the onset of symptoms, weight in kg, height in meter combined to report BMI in kg/m^2, Charlson score, Use of adjuvant oxygen, Lung CT-Scan results : extent of lesion <25%/25-50%/50-75%/>75%, Lymphocytes, platelet, CRP count at the time of diagnosis and 7 days after, GFR at diagnosis ml/min /1.73m2, ABO group, Rhesus antibody, Nasopharyngeal RT PCR initial Cycle Threshold

CONTACTS AND LOCATIONS:
Locations (1):
- Service SSR Gériatrique, Strasbourg, France